CLINICAL TRIAL: NCT01044199
Title: A Single Center, Open-Label, Study of Intradermal Administration of an Inactivated PCEC Rabies Vaccine in Adult Subjects
Brief Title: Study of Intradermal Administration of PCEC Rabies Vaccine
Acronym: Rabies-ID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCEZID-5506; IND-13814 (Other: CDC); CDC-IRB 5506 (Other: CDC)
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Rabies Prevention; Rabies Exposure
Keywords: rabies; rabies vaccine; purified cultured embryo chicken rabies vaccine
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1: Pre-EP ID (Experimental): Group of participants receiving PCEC rabies vaccine intradermally with the Pre-Exposure schedule.
  Interventions: Biological: PCEC rabies vaccine given intradermally
- 2: Pre-EP IM (Active Comparator): Group of participants receiving PCEC rabies vaccine intramuscular with the Pre-Exposure schedule.
  Interventions: Biological: PCEC rabies vaccine administered intramuscularly
- 3: Booster ID (Experimental): Group of participants receiving PCEC rabies vaccine intradermally with the Booster schedule.
  Interventions: Biological: PCEC rabies vaccine given intradermally
- 4: Booster IM (Active Comparator): Group of participants receiving PCEC rabies vaccine intramuscular with the Booster schedule.
  Interventions: Biological: PCEC rabies vaccine administered intramuscularly

INTERVENTIONS:
Biological: PCEC rabies vaccine given intradermally — PCEC rabies vaccine will be given intradermally compared with intramuscular administration (standard), in 2 different schedules: Pre-Exposure schedule for participants never vaccinated against rabies before; and Booster schedule for participants vaccinated against rabies in the past.
  Other Names: RabAvert
  Arms: 1: Pre-EP ID; 3: Booster ID
Biological: PCEC rabies vaccine administered intramuscularly — PCEC rabies vaccine will be given intradermally compared with intramuscular administration (standard), in 2 different schedules: Pre-Exposure schedule for participants never vaccinated against rabies before; and Booster schedule for participants vaccinated against rabies in the past.
  Other Names: RabAvert
  Arms: 2: Pre-EP IM; 4: Booster IM

SUMMARY:
The purpose of this study is to determine immunogenicity and safety of intradermal administration of the PCEC rabies vaccine in adults.

DETAILED DESCRIPTION:
Approximately 16,000-39,000 persons come in contact with potentially rabid animals and receive rabies postexposure prophylaxis (PEP) each year in the US. To appropriately manage potential human exposures to rabies, the risk for infection must be accurately assessed. Administration of rabies PEP is a medical urgency, not a medical emergency, but decisions must not be delayed. Prophylaxis is occasionally complicated by adverse reactions, but these reactions are rarely severe. Current data on the safety and efficacy of active and passive rabies vaccination were derived from both human and animal studies. Timely and appropriate human pre-exposure prophylaxis (Pre-EP) and PEP will prevent human rabies. Currently in the US, the approved dosage and administration for PEP in previously unvaccinated persons consists of the administration of vaccine (HDCV or PCECV) and HRIG. Vaccine is administered IM on days 0, 3, 7, 21, and 28 (deltoid area). The approved dosage and administration for pre-exposure prophylaxis (Pre-EP) consists of three 1.0-mL injections of vaccine (HDCV or PCECV) administered IM (deltoid area), one injection per day on days 0, 7, and 21 or 28). Intradermal (ID) route of administration of rabies vaccination is used in certain countries both for PEP and Pre-EP, and approved by WHO for modern potent cell culture vaccines. Recent studies outside the USA found the use of PCEC rabies vaccine by ID administration immunogenic and safe.

The primary goals of this study are to obtain additional safety and immunogenicity data on ID administration of 0.1 mL doses of the inactivated PCEC rabies virus vaccine in adults. Given the need to provide alternative routes of administration to the current approved intramuscular route in order to protect a larger number of people facing potential vaccine shortages. The data yielded by this clinical trial will provide evidence to support alternative route of administration and dose of PCECV in the US.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory personnel, epidemiologists, EISOs, veterinary students, interns, and other first responders at CDC; other CDC employees; and healthy volunteer adults. Persons who contact the study coordinator will be assessed for possible occupational exposure to rabies using the risk assessment form (appendix E). The volunteers reporting occupational exposure will be selected to enter the study.
2. Male or nonpregnant females (as indicated by a negative urine pregnancy test prior to first dose of vaccine), aged 18 years and older.
3. Women of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (i.e., barrier method, abstinence, or licensed hormonal methods) for the entire study period.
4. Be in good health, as determined by vital signs (pulse, blood pressure, oral temperature), medical history, and a targeted physical examination based on medical history.
5. Able to understand and comply with planned study procedures.
6. Provide informed consent prior to any study procedures and be available for all study visits.
7. Have health insurance.

Exclusion Criteria:

1. Have a known allergy to PCECV.
2. Have a known allergy or sensitivity to eggs or latex (in the stopper).
3. Have a positive urine pregnancy test prior to first vaccine dose (female of childbearing potential age).
4. Are immunosuppressed as a result of an underlying illness or treatment.
5. Have active neoplastic disease or a history of any hematologic malignancy.
6. Are using oral or parenteral steroids, high-dose inhaled steroids (>800 μg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs.
7. Have a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
8. Have an acute illness that is accompanied by an oral temperature greater than 100.4°F, within 1 week of vaccination.
9. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during the 1st month of the study period.
10. Have any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
11. He/she is a CDC worker under direct supervision of any of the primary study investigators (Dr. Sergio Recuenco, and Dr. Eli Warnock).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have virus-neutralizing antibody titers of at least 1:5 serum dilution by the RFFIT, 14 days after receipt of the last dose of the vaccine. | 14 days after receipt of the last dose of the vaccine.
Adverse event (AE) or serious adverse event (SAE) information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessment). | Imnediately after fisrt dose to completion of the study 6 months later.

SECONDARY OUTCOMES:
Proportion of subjects who have virus-neutralizing antibody titers of at least 1:5 serum dilution by the RFFIT in each group. | 14, 60, 120 and 160 days after last dose of vaccine.
Distribution GMTs of virus-neutralizing antibody titers in each group. | 14, 60, 120 and 160 after last dose of vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Recuenco, MD,MPH,DrPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- CDC Occupational Clinic, Atlanta, Georgia, United States